CLINICAL TRIAL: NCT01276574
Title: Epithelial Ovarian Cancer- Staging and Response to Chemotherapy Evaluated by PET/CT(positron Emission Tomography/computed Tomography)
Brief Title: Epithelial Ovarian Cancer- Staging and Response to Chemotherapy Evaluated by PET/CT
Acronym: Mupet
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 53/180/2009
Record Dates: First submitted 2010-09-01; First posted 2011-01-13 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: PET/CT; Ovarian cancer; HE4
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumour samples, whole blood and serum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine, whether there is clinical benefit of using fdg-PET/CT (F-18-fluorodeoxyglucose- positron emission tomography/computed tomography)compared to contrast-enhanced CT in primary treatment of advanced epithelial ovarian cancer (EOC)

* Objectives

  * the impact of preoperative PET/CT compared to CT on EOC stage definition
  * to compare the value of preoperative PET/CT, CT and laparoscopy in intra-abdominal tumour assessment. Laparotomy findings evaluated by surgeon and histopathologic results serve as the reference standard.
  * to compare serum markers HE4(human epididymis protein 4) and CA125 (cancer antigen 125) with FDG-PET/CT and CT in treatment response evaluation during neoadjuvant chemotherapy and primary treatment of EOC
  * to compare FDG PET/CT based treatment response evaluation with RECIST and GCIG criteria
* Methods

  * All the patients will undergo FDG-PET/CT prior surgery, after possible neoadjuvant chemotherapy (NACT) and 4 weeks after completion of primary platinum-based chemotherapy.
  * CA125 and HE4 levels are measured pre-operatively, with every chemotherapy cycle and regularly during follow-up until 1st disease relapse

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with advanced epithelial ovarian, primary peritoneal cancer or fallopian tube cancer.
* age 18-79 years
* informed concent

Exclusion Criteria:

* diabetes (for PET/CT analyses)
* previous cancer

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical suspicion of advanced EOC referred to surgery to Turku University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-10; Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PET/CT (positron emission tomography/computed tomography)compared with contrast-enhanced CT in preoperative evaluation of disease burden in patients with advanced Epithelial ovarian cancer (EOC). | PET/CT, contrast-enhanced CT and surgical status and histopathological findings are compared 1 month after surgery
  Patient is scanned with whole body Fdg PET/CT and contrast-enhanced CT in a row within 3 weeks preoperatively. Findings are compared with intraoperative surgical status evaluated by operator and confirmed with biopsies.

SECONDARY OUTCOMES:
Neoadjuvant chemotherapy (NACT) response evaluation with PET/CT compared with contrast-enhanced CT after 3 cycles of chemotherapy | Outcome measure: after interval debulking surgery, about 4 months
  Fdg PET/CT and a contrast-enhanced CT are performed in a row at the time of diagnosis and repeated after 3 cycles of chemotherapy. Finding are compared with disease status in the interval debulking surgery evaluated by operator and histological specimen.
Serial measurement of HE4 (human epididymis protein 4) and CA125 (cancer antigen 125)during primary treatment of EOC (Epithelial ovarian cancer) | From diagnosis until the end of EOC primary therapy, about 8 months
  HE4 and CA125 are measured at the time of diagnosis, perioperatively, and at each chemotherapy cycle (6-9). Treatment outcome is evaluated with contrast-enhanced CT at the end of primary therapy. HE4 and CA125 are compared with each other in different treatment outcomes (complete response, partial response, stable disease and progression) and PFS and OS
Response to first line treatment: evaluation with PET/CT | PET/CT taken about 4 weeks after the last chemotherapy cycle
  Treatment outcome measured with RECIST 1.1 and GCIG criteria is compared with PET/CT results. The prognostic role of persistent metabolic activity in PET/CT is evaluated.
HE4 and CA125 in 1st relapse | Long time follow up ad 10 years
  Prognostic value of HE4 and CA125 at 1st recurrence (defined with RECIST1.1. and GCIG criteria) is evaluated against post progression survival

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Hynninen, Adj prof, Study Director — Turku University hospital, Department of Obstetrics and Gynecology; Johanna Hynninen, MD, PhD, Principal Investigator — Turku University hospital, Department of Obstetrics and Gynecology
Locations (1):
- Turku University hospital, Turku, Finland

REFERENCES:
- [Derived] Salminen L, Gidwani K, Grenman S, Carpen O, Hietanen S, Pettersson K, Huhtinen K, Hynninen J. HE4 in the evaluation of tumor load and prognostic stratification of high grade serous ovarian carcinoma. Acta Oncol. 2020 Dec;59(12):1461-1468. doi: 10.1080/0284186X.2020.1827157. Epub 2020 Oct 8. PMID 33030975
- [Derived] Laasik M, Kemppainen J, Auranen A, Hietanen S, Grenman S, Seppanen M, Hynninen J. Behavior of FDG-avid supradiaphragmatic lymph nodes in PET/CT throughout primary therapy in advanced serous epithelial ovarian cancer: a prospective study. Cancer Imaging. 2019 May 29;19(1):27. doi: 10.1186/s40644-019-0215-7. PMID 31142357
- [Derived] Hynninen J, Kemppainen J, Lavonius M, Virtanen J, Matomaki J, Oksa S, Carpen O, Grenman S, Seppanen M, Auranen A. A prospective comparison of integrated FDG-PET/contrast-enhanced CT and contrast-enhanced CT for pretreatment imaging of advanced epithelial ovarian cancer. Gynecol Oncol. 2013 Nov;131(2):389-94. doi: 10.1016/j.ygyno.2013.08.023. Epub 2013 Aug 29. PMID 23994535
- [Derived] Hynninen J, Lavonius M, Oksa S, Grenman S, Carpen O, Auranen A. Is perioperative visual estimation of intra-abdominal tumor spread reliable in ovarian cancer surgery after neoadjuvant chemotherapy? Gynecol Oncol. 2013 Feb;128(2):229-32. doi: 10.1016/j.ygyno.2012.11.007. Epub 2012 Nov 9. PMID 23142076
- [Derived] Hynninen J, Auranen A, Carpen O, Dean K, Seppanen M, Kemppainen J, Lavonius M, Lisinen I, Virtanen J, Grenman S. FDG PET/CT in staging of advanced epithelial ovarian cancer: frequency of supradiaphragmatic lymph node metastasis challenges the traditional pattern of disease spread. Gynecol Oncol. 2012 Jul;126(1):64-8. doi: 10.1016/j.ygyno.2012.04.023. Epub 2012 Apr 24. PMID 22542580